CLINICAL TRIAL: NCT06375369
Title: Adoption and Enhancement of a Care Pathway for Children With Medical Complexity: an Implementation Evaluation Project for Tracheostomy in Pediatrics
Brief Title: Digital Health Pathway for Children With Medical Complexity Requiring Tracheostomy
Acronym: DECIDE-T
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00127121
Record Dates: First submitted 2024-04-13; First posted 2024-04-19 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Tracheostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-implementation (No Intervention): Subjects undergoing tracheostomy procedure before the implementation of DECIDE-T
- Post-implementation/Intervention (Active Comparator): Subjects undergoing tracheostomy procedure after the implementation of DECIDE-T
  Interventions: Procedure: Digital health pathway for children with medical complexity requiring tracheostomy (DECIDE-T)

INTERVENTIONS:
Procedure: Digital health pathway for children with medical complexity requiring tracheostomy (DECIDE-T) — The intervention involves developing a standardized clinical pathway for these children requiring tracheostomy. The pathway comprises of a hospital to home directive, incorporating digital health solutions to support family, caregivers, and healthcare professionals. These digital supports include but are not limited to a Connect Care pathway, resources to aid families to make informed choices during the clinical decision-making process, education modules and high-fidelity simulations to enhance family/caregiver education, an online parental resource center and access to peer support (spanning from hospital to community) and a telehealth post discharge program.
  Arms: Post-implementation/Intervention

SUMMARY:
The DECIDE-T project is developing a standardized clinical pathway specifically for pediatric patients who require tracheostomy with or without long-term ventilation (tracheostomy/LTV). These patients represent a small portion of Alberta's population but account for over 50% of pediatric patients hospitalized for more than 180 days. The pathway will include a hospital-to-home directive that incorporates digital health solutions to provide support to families, caregivers, and healthcare professionals. Digital supports will include a Connect Care pathway, resources for informed decision-making, educational modules, high-fidelity simulations for family and caregiver education, an online parental resource center, and access to peer support within the hospital and community, as well as a post-discharge telehealth program.

The goal of the DECIDE-T project is to reduce hospital stays and associated costs for children requiring tracheostomy/LTV, as well as to decrease mental distress and burnout experienced by their caregivers and families.

DETAILED DESCRIPTION:
BACKGROUND: Medical advances have resulted in more children surviving critical illness and then living with medical complexity. Children discharged after critical illness with a tracheostomy-a surgical opening created through the neck to form an artificial airway that can be used for mechanical ventilation-are an example of this medically complex, technologically-dependent patient population. In Alberta, care for these children is centralized at the Stollery and Alberta Children's Hospitals. Fewer than 40 tracheostomized patients/year account for >50% of pediatric patients hospitalized for over 180 days and average $484.660/patient/year-more than 30% of Alberta's annual pediatric acute care budget. These tertiary centers, however, lack a provincial standardized tracheostomy care pathway and, based on current guidelines, have substantial variations in practice, program inefficiencies, and barriers to care. This causes: 1) compromised health and disease burden for patients; 2) inconsistent and poorly informed decision-making; 3) increased stay in intensive care and hospital; 4) systemic inequities for certain subpopulations; and 5) substantial burdens for families-caregivers and healthcare providers (HCPs), causing burnout and long-lasting mental health complications. These factors result in a high cost for the health system and potential detriment to the care of other pediatric patients.

DIGITAL SOLUTION: Investigators propose the adaptation, implementation, and assessment of a provincial Digital hEalth Pathway for ChIldren with MeDical ComplExity requiring Tracheostomy/LTV (DECIDE-T). The DECIDE-T model will comprise a hospital-to-home journey, education and peer support digital solutions and a telemedicine follow-up program to support families-caregivers and HCPs looking after tracheostomized children.

PRIMARY OBJECTIVE: Reduce hospital stay and costs by 40%; SECONDARY OBJECTIVE: decrease families-caregivers mental stress and HCPs moral distress using validated measures.

APPROACHES: The key components of DECIDE-T will be defined using evidence-based guidelines and consultation with families-caregivers, HCPs, and other stakeholders. Scientific methods will be used to evaluate outcomes after implementation of DECIDE-T.

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years
* First tracheostomy placement

Exclusion Criteria:

-

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospital length of stay | 12 months
  The total duration of patient stay in hospital
ICU length of stay | 12 months
  The total duration of patient stay in ICU
ICU readmission | 12 months
  Rate of ICU re-admissions during the index hospitalization
Mortality | 12 months
  All cause mortality during admission
Decannulation | 12 months
  Successful decannulation during admission
Duration of tracheostomy | 12 months
  Time between tracheostomy placement and successful decannulation
Tracheostomy adverse events | 12 months
  Tracheostomy related adverse events during admission
Hospital cost | 12 months
  Total cost of hospital stay
Hospital readmission | 12 months
  Rate of hospital re-admissions after index hospital discharge
Net-monetary benefit of DECIDE-T | 12 months
  The healthcare cost-savings attributable to DECIDE-T as the difference between the mean cost per index admission for patients treated before and after DECIDE-T implementation. The costs will include costs of hospitalizations, outpatient visits, physician claims, home care costs where available, readmissions after index discharge

SECONDARY OUTCOMES:
Caregivers mental stress | 12 months
  The mental distress and burnout of caregivers/families of children requiring tracheostomy using the Pediatric Inventory for Parents (PIP). The PIP is a questionnaire comprising 42 items, grouped into four domains or subscales (Communication (CM), Emotional Distress (ED), Medical Care (MC), and Role Function (RF)). Its purpose is to measure the levels of stress suffered by parents caring for a child with a chronic illness or requires prolonged medical monitoring. Responses are provided using a five-point Likert scale, ranging from 1 ("never/not at all") to 5 ("very often/extremely"). Higher scores indicate higher levels of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Castro Codesal, MD, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No